CLINICAL TRIAL: NCT02375191
Title: A Comparative Study of the Effect of Epidural Dexmedetomidine Versus Fentanyl Added to Ropivacaine in Pediatric Orthopedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2014-0921
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Congenital Skelectal Anomaly
MeSH Terms: interventions — Fentanyl; Dexmedetomidine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fentanyl (Active Comparator): 0.2% ropivacaine+ 1 mcg/kg fentanyl
  Interventions: Drug: fentanyl; Drug: Ropivacaine
- dexmedetomidine (Experimental): 0.2% ropivacaine+1 mcg/kg dexmedetomidine
  Interventions: Drug: dexmedetomidine; Drug: Ropivacaine

INTERVENTIONS:
Drug: fentanyl
  Arms: fentanyl
Drug: dexmedetomidine
  Arms: dexmedetomidine
Drug: Ropivacaine

SUMMARY:
The purpose of this study is to evaluate the effect of epidural dexmedetomidine added to ropivacaine in pediatric orthopedic surgery

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients aged from 3 to 12 years undergoing orthopedic mechanical correction surgery

Exclusion Criteria:

* coagulopathy, refusal (parents), current infection on the lumbar area, spinal tract pathology

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score | During 48 hrs after pediatric orthopedic surgery
  CHEOPS, FLACC score were measured

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, Seoul, South Korea